CLINICAL TRIAL: NCT05020418
Title: Promoting De-Implementation of Inappropriate Antimicrobial Use Following Cardiac Device Procedures
Brief Title: De-Implementation of Inappropriate Antimicrobial Use After Cardiac Device Procedures
Acronym: CIED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Westyn Branch-Elliman, Assistant Professor of Medicine, VA Boston Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB 1585926
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Antibiotics Causing Adverse Effects in Therapeutic Use
Keywords: cardiac devices; antimicrobial use; chart review; learning/unlearning; de-implementation; de-adoption; Hybrid III implementation trial; antimicrobial stewardship; peri-operative antimicrobial use; peri-procedural antimicrobial use; peri-procedural infection control; stepped-wedge

STUDY DESIGN:
Intervention Model Description: Cardiac device procedures performed within the national VA healthcare system during the period from Fiscal Year (FY) 16-24 will be identified using a list of relevant Current Procedural Terminology (CPT) codes. Based on our preliminary results, we anticipate that the VA Corporate Data Warehouse (CDW) EP Procedures Cohort (electronic surveillance cohort) will include approximately 100,000 cardiac device cases. Because this cohort is based in CDW, once a Veteran undergoing a device procedure is identified using CPT codes, the orders, procedures, and consults that occurred during the 90-day window following the procedure can be extracted from the VA Electronic Health Record (EHR) In addition to the full cohort, the implementation bundle will be tested at the three high-volume intervention sites (~1500 cases per year). Roll out of the interventions will occur in a stepped manner, such that pre- and post- intervention data will be collected at all sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Device Cohort (Experimental): This study is open to any adult VA patient with data about a cardiac device procedure performed in the electrophysiology laboratory entered into the national VA EHR. During FY 20-FY 24, we anticipate that this will include approximately 9,000 patients per year, or a total of 50,000 patients. In addition, cases that were previously accessed and used to develop the infection monitoring system, and the quality metric monitoring system, may also be included. This includes all patients entered in the VA Clinical Assessment Reporting and Tracking - Electrophysiology Cohort (CART-EP) database during the period from 2006-2016, and all VA patients who received a cardiac device procedure during the period from 2010-2019. This includes another approximately 50,000 patients, for a total of 100,000 patients.
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — Intervention sites will receive a multi-faceted implementation intervention, which will include external and internal blended facilitation, education materials for providers and patients, and audit and feedback about practices and outcomes with benchmarking to non-intervention sites.

SUMMARY:
This project will use automated audit and feedback to improve compliance with antimicrobial prophylaxis guidelines for CIED procedures that we anticipate will translate into better outcomes for our patients. A multi-faceted implementation bundle to promote de-implementation of guideline discordant care will be tested at three intervention sites. Materials and tools will then be disseminated throughout the VA healthcare system if the intervention is found to be effective.

DETAILED DESCRIPTION:
Aim I tests the hypothesis that a multi-faceted implementation strategy that includes educational sessions with members of electrophysiology teams and locally-adapted monthly surveillance reports about guideline-concordant pre-procedural antimicrobial use and guideline-discordant post-procedural antimicrobial use, 90-day incidence of CIED infections, and 90-day incidence of C. difficile infections and 7-day incidence of AKI that will be delivered to local infectious diseases champions and shared with electrophysiology teams using blended facilitation will promote uptake of best practices and improve outcomes. This hypothesis incorporates learning/unlearning and fills a major gap caused by the dearth of rigorous de- implementation and de-adoption studies. Aim II tests the hypothesis that electronic health records (EHRs) and medical informatics have advanced to the point that it will be feasible, during the next four years, to establish an audit and feedback surveillance system that can be scaled and disseminated widely across the VA.

This study will use mixed qualitative and quantitative methods to address the study aims. This will include interviews with key stakeholders and quantitative measurement of quality metrics (e.g., pre-and post-procedure antimicrobial use) and outcomes (e.g., cardiac device infections, acute kidney injuries, C. difficile infections).

All patients receiving a cardiac device implantation within the VA healthcare system during the study period may be potentially included. Medical records previously reviewed and accessed may also be included for validation, testing, and optimization of electronic algorithms. In addition to the VA patients who will participate, key stakeholders for infection prevention in the cardiac device laboratory (e.g., providers, nurses, electrophysiology laboratory staff) will also participate in interviews. Active implementation will occur at 3 VA sites, a passive dissemination process will occur at all VA sites with a cardiac device laboratory (~78 VA sites).

High quality studies establish that prolonged prophylaxis has no beneficial impact on CIED-related infection rates but worsens outcomes and leads to preventable deaths. Despite guidelines specifically recommending against prolonged prophylaxis, this practice is common in cardiac electrophysiology laboratories, including VA and non-VA hospitals. At the same time, antimicrobial resistance and overuse represent critical threats to the health of the population. This intersection- inappropriate prescribing and a critical need to improve use-- creates an urgent need for research into methods to promote adoption of best antimicrobial use and de-implementation of ineffective and harmful prescribing. IT-based solutions for improving antimicrobial use, including antimicrobial prophylaxis, is a quality-improvement strategy endorsed by The Joint Commission. This project will advance this concept and couple learning/unlearning processes to promote uptake of best practices. If effective, this model can be replicated in other settings of care to improve antimicrobial use.

ELIGIBILITY:
Inclusion Criteria:

* This study is open to any adult VA patient with data about a cardiac device procedure performed in the electrophysiology laboratory entered into the national VA EHR.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
cardiac device infection | 90 days
  Incidence of cardiac device infections
C. difficile infections | 90 days
  Incidence of C. difficile infections
Acute Kidney Injury (AKI) | 7 days
  Incidence of AKI
Pre-procedure Antimicrobial Use | 1 day
  Proportion of cases with guideline-concordant pre-procedure antimicrobial use defined as appropriate antimicrobials administered within 1 hour prior to incision.
Post-procedure Antimicrobial Use | 14 days
  Proportion of cases with guideline-concordant post-procedure antimicrobial use defined as antibiotics administered for prevention of cardiac device infection (not for pre-existing infection) lasting for greater than 24 hours following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Westyn Branch-Elliman, MD, Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
A de-identified, anonymized dataset will be created and shared upon request and executing a Data Use Agreement (DUA) following VA research regulations, current guidance can be found in Veteran's Health Administration (VHA) Directive 1080.01(1) last updated March 2021.

REFERENCES:
- [Derived] Branch-Elliman W, Lamkin R, Shin M, Mull HJ, Epshtein I, Golenbock S, Schweizer ML, Colborn K, Rove J, Strymish JM, Drekonja D, Rodriguez-Barradas MC, Xu TH, Elwy AR. Promoting de-implementation of inappropriate antimicrobial use in cardiac device procedures by expanding audit and feedback: protocol for hybrid III type effectiveness/implementation quasi-experimental study. Implement Sci. 2022 Jan 29;17(1):12. doi: 10.1186/s13012-022-01186-8. PMID 35093104